CLINICAL TRIAL: NCT04740021
Title: A Single-arm, Open-lable, Multicenter, Phase II Clinical Study of LP002 in Combination With Chemotherapy for Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Study of LP002 in Combination With Chemotherapy for Patients With Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou HoudeAoke Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP002-II-SCLC-01
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: LP002+EP (Experimental): Participants recieve LP002 10 mg/kg intravenous (IV) on day 1 PLUS carboplatin titrated to an area under the plasma drug concentration-time curve [AUC] 5 IV on day 1 PLUS etoposide 100 mg/m^2 IV on days 1, 2 and 3 of each 21-day cycle
  Interventions: Drug: LP002; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: LP002 — 10 mg/kg administered as IV infusion on Day 1 of each 21-day cycle.
Drug: Carboplatin — AUC 5 administered as IV infusion on Day 1 of each 21-day cycle.
Drug: Etoposide — 100 mg/m^2 administered as IV infusion on Day 1, 2 and 3 of each 21-day cycle.

SUMMARY:
LP002 is a highly selected recombinant humanized anti-PD-L1 monoclonal antibody. This is a single-arm, multicenter study to evaluate the efficacy and safety of LP002 in combination with chemotherapy in patients with extensive stage samll cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial;
* Age ≥ 18 and ≤ 79 years old, male or female;
* Histologically or cytologically diagnosed with ES-SCLC (according to the Veterans Administration Lung Study Group staging system).
* No prior systemic therapy for ES-SCLC.
* Patients who have received prior chemoradiotherapy for limited-stage SCLC must have been treated with curative intent and experienced a treatment-free interval of at least 6 months since last chemotherapy, radiotherapy, or chemoradiotherapy cycle from diagnosis of extensive-stage SCLC.
* Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Has a life expectancy of ≥3 months.
* Has at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Has adequate organ function.
* Female participants of childbearing potential should have a negative pregnancy within 72 hours before the first dose of trial treatment. Male and female participants should agree to use an adequate method of contraception during the experiment and 24 weeks after the last administration of the test drugs.

Exclusion Criteria:

* Histologically or cytologically confirmed mixed SCLC.
* Suffered from other malignant tumors in the past 5 years (except skin basal cell carcinoma, squamous cell carcinoma, and cervical carcinoma in situ that have been effectively controlled).
* Prior to the first administration of the study drug, there was a grade > 1 toxicity (excluding hair loss) caused by previous anti-tumor treatments.
* Has received prior therapy with an anti-PD-1, or anti-PD-L1, or anti-CTLA-4 agents.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Uncontrolled or symptomatic hypercalcemia.
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≤ 1 week prior to the first dose of trial treatment.
* Has active autoimmune disease that has required systemic treatment in past 2 years.
* Has received a major surgery within 4 weeks prior to the first dose of trial treatment.
* Has received system treatment with corticosteroids (dose >10mg/day prednison or other therapeutic hormones) within 2 weeks prior to the first dose of trial treatment.
* Previous or present interstitial lung disease or non-communicable pneumonia, except for radiation pneumonia.
* Has uncontrolled systemic disease, such as diabetes or hypertension.
* Has a history of testing positive for human immunodeficiency virus (HIV), or known acquired immunodeficiency syndrome (AIDS), or stem cell transplantation or organ transplantation.
* Has untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 500 IU/ mL or active hepatitis C virus (HCV). Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA < 10^3 copies/ml or <500 IU/ mL) , and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
* Has serious infections within 4 weeks or active infections requiring systemic treatment within 2 weeks prior to the first dose of trial treatment.
* Has a history of severe allergic reaction to any other monoclonal antibodies.
* Has participated in other anticancer drug clinical trials within 4 weeks.
* Is pregnant or breastfeeding.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 15 months
  PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 assessed by investigators or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to approximately 15 months
  ORR was defined as the percentage of participants who have a complete response (CR) or a partial response (PR), per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigators.
Disease Control Rate (DCR) | up to approximately 15 months
  DCR was defined as the percentage of participants who have a CR or a PR or a stable disease (SD), per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigators.
Duration of Response (DOR) | up to approximately 15 months
  DOR was defined as the time from the first documented evidence of a response of CR or PR, per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigators.
Number of Participants Who Experienced an Adverse Event (AE) | up to approximately 15 months
  An adverse event was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which did not necessarily have to have had a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Affiliated Hospital Of Jiangnan University, Wuxi, Jiangsu
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Xinjiang Medical University Cancer Center, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan